CLINICAL TRIAL: NCT03794167
Title: Randomized Phase II Multi-center Trial of Busulfan, Etoposide, and Cyclophosphamide Versus Busulfan, Etoposide, and Melphalan as Conditioning Therapy for Autologous Stem-cell Transplantation(ASCT) in Patients With Non-Hodgkin's Lymphoma
Brief Title: BuCE Versus BuME as Conditioning Therapy in Non-Hodgkin's Lymphoma
Acronym: CISL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Soonchunhyang University Hospital (Other)
Responsible Party: Principal Investigator, Jong-Ho Won, Professor, Soonchunhyang University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CISL 12-05
Record Dates: First submitted 2019-01-03; First posted 2019-01-04 (Actual); Last update posted 2019-01-07 (Actual); Status verified 2019-01

CONDITIONS: Non-hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Busulfan; Cyclophosphamide; Etoposide; Melphalan

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- busulfan cyclophosphamide etoposide (Experimental): busulfan 3.2 mg/kg/day i.v. on days -8,-7, and -6, cyclophosphamide 50mg/kg/day i.v. on days -3 and -2 etoposide 400mg/m2 day i.v. on days -5 and -4
  Interventions: Drug: Busulfan; Drug: Cyclophosphamide; Drug: Etoposide
- busulfan melphalan etoposide (Active Comparator): busulfan 3.2 mg/kg/day i.v. on days -8,-7, and -6 melphalan 50mg/m2/day i.v. on days -3 and -2 etoposide 400mg/m2 day i.v. on days -5 and -4
  Interventions: Drug: Busulfan; Drug: Etoposide; Drug: Melphalan

INTERVENTIONS:
Drug: Busulfan — busulfan 3.2 mg/kg/day i.v. on days -8,-7, and -6
  Other Names: Busulfex
Drug: Cyclophosphamide — cyclophosphamide 50mg/kg/day i.v. on days -3 and -2
  Arms: busulfan cyclophosphamide etoposide
Drug: Etoposide — etoposide 400mg/m2 day i.v. on days -5 and -4
Drug: Melphalan — melphalan 50mg/m2/day i.v. on days -3 and -2
  Other Names: Alkeran
  Arms: busulfan melphalan etoposide

SUMMARY:
The investigators developed a protocol comparing busulfan/cyclophosphamide/etoposide (BuCE) and busulfan/melphalan/etoposide (BuME) regimen as a conditioning for high-dose therapy (HDT) in the patients with high risk or relapsed Non-Hodgkin's Lymphoma (NHL).

DETAILED DESCRIPTION:
Intravenous busulfan containing regimens as conditioning regimen have been used for both allogeneic and autologous stem cell transplantation in patients with hematologic and non-hematologic malignancies.

The investigators have previously studied that conditioning regimen of i.v. busulfan/melphalan/etoposide (BuME) was well tolerated and effective in patients with relapsed or high risk NHL. And busulfan/cyclophosphamide/etoposide (BuCE) conditioning regimen has been extensively utilized in ASCT for NHL.

Therefore, based on the encouraging results, the investigators will conduct a randomized phase II multicenter trial of BuCE versus BuME as conditioning therapy for ASCT in patients with NHL.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed aggressive NHL
2. Mantle cell lymphoma
3. salvage chemotherapy sensitive relapse/refractory NHL or high risk NHL with remission in induction chemotherapy
4. Performance status: Eastern Cooperative Oncology Group (ECOG) 0-2.
5. Age; 18-65
6. Adequate renal function: serum creatinine ≤ 1.5mg/dL
7. Adequate liver functions: Transaminase (AST/ALT) < 3 X upper normal value & Bilirubin < 2 X upper normal value

Exclusion Criteria:

1. low grade NHL
2. Any other malignancies within the past 5 years except curatively treated non-melanoma skin cancer or in situ carcinoma of cervix uteri
3. Other serious illness or medical conditions

   * Unstable cardiac disease despite treatment, myocardial infarction within 6 months prior to study entry
   * History of significant neurological or psychiatric disorders
   * Active uncontrolled infection (viral, bacterial or fungal infection)
4. Pregnant or lactating women, women of childbearing potential not employing adequate contraception
5. HIV (+)
6. Patients who have hepatitis B virus (HBV) (+) are eligible. However, primary prophylaxis using antiviral agents (i.e. lamivudine) is recommended for HBV carrier to prevent HBV reactivation during whole treatment period -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2012-06-01 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Rate of progression free survival | 2 years
  calculate from the date of ASCT until the time of disease progression, relapse, or death calculate from the date of ASCT until the time of disease progression, relapse, or death calculate from the date of ASCT until the time of disease progression, relapse, or death Calculate from the date of ASCT (autologous stem cell transplantation) until the time of disease progression, relapse, or death

SECONDARY OUTCOMES:
Rate of overall survival | 2 years
  calculate from the date of ASCT until the time of death from any causes
Rate of regimen related toxicity | 6 months
  calculate toxicities frequency

CONTACTS AND LOCATIONS:
Overall Officials: Jong-Ho Won, Professor, Principal Investigator — Soonchunhyang University Hospital
Locations (1):
- Jong-Ho Won, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No